CLINICAL TRIAL: NCT05176106
Title: Advancing the Health of Rural Communities in Uganda Through Strong Community Health Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015042
Record Dates: First submitted 2021-11-01; First posted 2022-01-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Incentives; Health Behavior; Health Care Utilization
Keywords: Community Health Workers; Incentives; Uganda; Motivation; Retention; Performance
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Parishes will be randomized to intervention or control. VHTs in the intervention parishes will receive the incentives package as part of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Randomized Parishes (Experimental): Parishes will be randomized in Masindi District to receive the intervention (i.e., an incentives package). VHTs who are active in that parish will thereby receive the incentives intervention.
  Interventions: Behavioral: CHW Incentives Intervention
- Control-Randomized Parishes (No Intervention): Non-intervention randomized parishes will be the control parishes. Active VHTs in the control parishes will not receive the incentives intervention.

INTERVENTIONS:
Behavioral: CHW Incentives Intervention — The intervention comprises of an incentives package provided to VHTs who are active in the intervention-randomized parishes. It will comprise of items that will motivate them and support their work as VHTs in the community.
  Arms: Intervention-Randomized Parishes

SUMMARY:
The overarching goal of this study is to improve the health of women and children in rural areas of Uganda through strengthening of the community health workforce, which provides critical health services to the rural poor.

DETAILED DESCRIPTION:
Uganda, like several countries in Sub-Saharan Africa, faces a shortage of skilled healthcare workers, and a disproportionate concentration of workers in urban areas. This disparity has dire consequences for rural populations, who have higher fertility rates, lower utilization of maternal and child health services, lower levels of access to safe drinking water and sanitation services, and poorer vaccination coverage. Women and children in rural and remote communities bear the disproportionate brunt of poor access to and poor quality of health care. Village Health Teams (VHTs), Uganda's community health workers (CHW), were introduced to address some of these inequities by providing basic health services to the rural poor. However, like many CHW programs globally, the VHT program has high levels of attrition, owing to inadequate systems and financial support.

The objectives of this study are to understand:

1. What structure and group of incentives is best suited to motivate VHTs, improve their performance in the delivery of services, and increase their retention in the health workforce?
2. What is the behavioral mechanisms through which new incentives may work or fail to work?
3. How do the changes in the national VHT program impact utilization of maternal and child health services, sanitary practices, and perception of quality of health services at the community-level? What is the impact of COVID-19 on VHT practices on community health?

This study will evaluate a 1-year incentives intervention provided to VHTs in Uganda's Masindi District. It is a two-armed clinical trial, where parishes will be randomized to the incentives intervention (i.e., an incentives package will be provided to VHTs practicing in the intervention parishes; control parishes VHTs will not receive an incentives package). The primary outcomes include assessing VHT performance, VHT motivation, VHT retention, trends in utilization of maternal and child health services, and trends in the adoption of sanitary practices. Outcomes for VHT performance, VHT retention, trends in utilization of maternal and child health services, and trends in adoption of sanitary practices will be measured monthly. Outcomes for VHT motivation will be measured twice, at baseline (Month 1) and endline (Month 12).

ELIGIBILITY:
Inclusion Criteria:

* Must be an active VHT in Uganda's Masindi district.

Exclusion Criteria:

* Anyone who fails to meet the inclusion criteria specified above will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in VHT Performance | Measured monthly for 12 months
  Measure change in average number of VHT visits made over the course of the 1-year intervention. Types of VHT visits include: average number of home visits, antenatal care visits, postnatal care visits, visits to support immunization of children, visits to talk about safe drinking water, visits to examine latrines and observe handwashing, and number of referrals made to the health facility over the last month.
Change in VHT Motivation | Baseline (Month 1) and Endline (Month 12)
  Measure the percentage of VHTs who have improved motivation during the course of the 1-year intervention through use of the Close-To-Community (CTC) Provider Motivational Indicator Scale, which measures satisfaction, organizational commitment, community commitment, and work conscientiousness.
Change in VHT Retention | Measured monthly for 12 months
  Measure the percentage of VHTs who report to the health facility over the course of the 1-year intervention.
Change in Maternal and Child Health Services Utilization | Measured monthly for 12 months
  Measure change in maternal and child health services utilization, which includes proportion of antenatal care coverage, proportion of immunization coverage, and proportion of children under 5 who have been visited by a VHT, over the course of the 1-year intervention.
Change in Adoption of Sanitary Practices | Measured monthly for 12 months
  Measure changes in the adoption of sanitary practices, which includes assessing the average number of households with latrines, improved latrines, handwashing facilities, safe drinking water, and are open defecation free over the course of the 1-year intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data. All data that will be shared will be at the aggregate-level so that any identifying information is not identifiable and does not place the participant at additional risk.

REFERENCES:
- [Derived] Agarwal S, Tweheyo R, Pandya S, Obuya E, Kiyomoto A, Mitra P, Schleiff M, Nagpal T, Macis M, Rutebemberwa E. Impact of a recognition package as an incentive to strengthen the motivation, performance, and retention of village health teams in Uganda: a study protocol for a cluster randomized controlled trial. Trials. 2023 Jun 23;24(1):428. doi: 10.1186/s13063-023-07426-6. PMID 37353798